CLINICAL TRIAL: NCT01199640
Title: A Phase 2a Magnetic Resonance Imaging Study of the Safety and Efficacy of MLN1202 in Patients in Multiple Sclerosis
Brief Title: Study of the Safety and Efficacy of MLN1202 in Patients in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Clinical Research Monitor, Millennium Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MLN120204-063
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — plozalizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN1202 (Experimental)
  Interventions: Drug: MLN1202

INTERVENTIONS:
Drug: MLN1202 — Patients received 5 intravenous (IV) infusions of the study drug. The first 3 infusions were administered at 15-day intervals, followed by 2 infusions at 30-day intervals. Patients were randomized to receive 1 of 2 doses of MLN1202 (4mg/kg or 8mg/kg).

SUMMARY:
This was a phase 2a study of MLN1202 to determine safety, tolerability and initial efficacy in patients with relapsing-remitting multiple sclerosis (RRMS). It was conducted in 2 dose cohorts enrolling a total of 50 patients. Efficacy was assessed by comparing the numbers of new gadolinium-enhancing brain lesions during the screening and treatment periods.

ELIGIBILITY:
Inclusion Criteria:

Each patient was to have met all of the following inclusion criteria to be enrolled in the study:

* 18 years of age or older
* Diagnosis of relapsing-remitting multiple sclerosis (RRMS)
* An Expanded Disability Status Score (EDCC) of 0 to 5.5, inclusive
* Be willing and able to comply with the protocol for the duration of the study period
* Be willing to use adequate "double-barrier" contraceptive methods for the duration of the study period
* If female, must be neither pregnant or breast-feeding
* Written informed consent
* To be enrolled in the treatment phase of the study each patient must have a total of at least 2 new gadolinium-diethylenetriamine pentaacetic acid (Gd)-enhancing lesions seen over the series of 3 pretreatment magnetic resonance imaging (MRI)s.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria were not to be enrolled in the study:

* Diagnosis of primary progressive multiple sclerosis (PPMS) or secondary progressive multiple sclerosis (SPMS)
* Received any investigational drug or experimental procedure within 3 months prior to study day 0
* If the patient has received disease-modifying treatments they must be discontinued prior to study day 0 as follows:

  1. Cyclophosphamide or mitoxantrone- 6 months prior
  2. Interferons, glatiramer acetate and azathioprine- 12 weeks prior
  3. Methotrexate, IV immunoglobulin, cyclosporin, plasma exchange or corticosteroids- 8 weeks prior
* Never have been exposed to Tysabri® (natalizumab)or any other VLA-4 (α4β1)antagonist
* Have an active infection or be considered to be at high risk for developing an infection
* Have a history of hepatitis B, C or human immunodeficiency virus (HIV)
* Have a chest X-ray within 6 months of study day 0 with clinically significant findings or abnormalities
* Have inadequate renal or hepatic function
* Have a known history of cancer, except for distant history (>10 years) of carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin
* Received any live, attenuated vaccinations within 30 days prior to study day 0
* Have a history of illicit drug or alcohol abuse within 5 years of study day 0
* Have a history of hypersensitivity to prior monoclonal antibody (mAb) treatment
* Have a history of allergy or sensitivity to Gd
* Have a history that would preclude serial MRI scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-05; Primary Completion 2007-07 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of MLN1202 in patients with relapsing-remitting multiple sclerosis (RRMS) | Day 61- Day 330
  Vital sign measurement, physical examinations, multiple sclerosis (MS) relapses, changes in expanded disability status scale (EDSS) scores and standard laboratory test results, as well as the incidence of adverse events and serious adverse events
To determine the efficacy of MLN1202 in patients with RRMS | Day 0- Day 180
  Comparing the mean number of new gadolinium-diethylenetriamine pentaacetic acid (Gd)-enhancing lesions on magnetic resonance imaging (MRI) scans during the pretreatment phase with the mean number of new Gd-enhancing lesions found during the treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.